CLINICAL TRIAL: NCT00000336
Title: Safety and Efficacy of Selegiline in Outpatient Treatment for Cocaine
Brief Title: Selegiline in Outpatient Treatment for Cocaine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-3-0010-1; Y01-3-0010-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 1996-01

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Selegiline

INTERVENTIONS:
Drug: Selegiline

SUMMARY:
The purpose of this study is to evaluate the efficacy and clinical safety of selegiline in the treatment of cocaine dependence and to assess neurotoxicity (Magnetic Resonance Imaging, MRI) post-hoc as a possible variable for future stratification in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Meets DSM-IV criteria for cocaine. Agreeable to conditions of study and signed informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nursing women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1995-01; Primary Completion 1996-02 (Actual); Study Completion 1996-03 (Actual)

PRIMARY OUTCOMES:
Urine toxicology for cocaine
Self reports of cocaine and other drug use and craving
Evidence of change in neurotoxicity based on choreoathetoid movement assessments

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States